CLINICAL TRIAL: NCT01773538
Title: Diagnosis of Covert/Minimal Hepatic Encephalopathy by Means of Continuous Reaction Time Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mette Munk Lauridsen (Other)
Collaborators: Region of Southern Denmark (Other); Odense University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Mette Munk Lauridsen, MD, Phd student, Esbjerg Hospital - University Hospital of Southern Denmark
Organization: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CHECRT
Record Dates: First submitted 2013-01-07; First posted 2013-01-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cirrhosis; Hepatic Encephalopathy
Keywords: quality of life
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy | interventions — Lactulose; Rifaximin; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti cHE treatment arm (Active Comparator): Of 150 included patients aprox. 44 regardless of CRT and PSE test outcome will be offered to enter randomisation and 3 months follow up. Half of 44 patients will receive both lactulose, rifaximin and branched chain aminoacids (Bramino) the other half placebo.
  Interventions: Drug: Lactulose and rifaximin; Dietary Supplement: Branched Chain amino acids
- Placebo arm (Placebo Comparator): The goal of this intervention is to investigate whether the CRT method can detect an expected treatment response after initiation of the 3 named drugs know to ameliorate HE symptoms including psychometric test results.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lactulose and rifaximin — 3 months treatment. lactulose 25 Ml x3 per day. Rifaximin (550 mg) x 2 per day.
  Arms: Anti cHE treatment arm
Dietary Supplement: Branched Chain amino acids — 30 grams of branched chain amino acids (Bramino) per day is given to the patients in the antiHE treatment arm along with lactulose and rifaximin.
  Arms: Anti cHE treatment arm
Other: Placebo — Patients in the placebo-arm receives both placebo-Bramino, placebo-lactulose and placebo-rifaximin.
  Arms: Placebo arm

SUMMARY:
The investigators wish to investigate how the Continuous Reaction Time (CRT) method can be used in the diagnosis and monitoring of covert hepatic encephalopathy (cHE)in patients with cirrhosis of the liver. The hypothesis is that the CRT method (duration 10-2 minutes) can serve as a tool in the diagnosis and monitoring of cHE and is an alternative to using the Portosystemic Encephalopathy Test (PSE)(duration 20-25 minutes).

DETAILED DESCRIPTION:
Objective: The aim of this project is to investigate whether continuous reaction time measurements (CRT) are suitable as a screening and monitoring tool for covert hepatic encephalopathy (c/mHE).

Method:

Sub-protocol 1: As a part of this PhD protocol 100 healthy individuals and 50 with chronic disease (not liver cirrhosis) will be tested using the CRT and PSE tests. This is to determine the normal range for the PSE test in the Danish population.

Sub-protocol 2: A total of 120 (aprox. 145 to adjust for drop outs) patients with liver cirrhosis from two Danish hospitals will be examined with both CRT and with the test that is the closest we get to a gold standard, namely portosystemic encephalopathy test (PSE). We wish to examine if the CRT test agrees with the PSE test, which may be to time consuming to perform in everyday clinical practice, and with quality of life scores (SF-36 and Sickness Impact Profile). The relationship between the CRT and PSE test and various blood tests and the Charlston co-morbidity score will also be examined.

Sub-protocol 3: Forty-four of the 120 included patients will, regardless of CRT test result, be randomized to treatment with lactulose, rifaximin and branched chain amino acids (BCAA) or placebo lactulose, rifaximin and BCAA. This is to evaluate whether the CRT method is able to detect a response to treatment, and see if changes in psychometric tests (PSE and CRT) are in accordance with quality of life scores and predicts subsequent development of overt hepatic encephalopathy.

Perspective: CRT method should, if it proves good enough, continue to be the Danish test of choice and hopefully be more widely used in our country. The validation of tests for the diagnosis of covert hepatic encephalopathy will give cirrhotic patients with covert hepatic encephalopathy and reduced quality of life the best opportunity to be diagnosed and offered appropriate treatment. If the CRT method is not able to identify a population that benefits from anti-encephalopathy treatment other screening and monitoring tests should be used.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteers:

* Age> 18 years
* Written informed consent
* Speak and understand Danish

For patients:

* Age > 18 years
* Liver cirrhosis confirmed by biopsy or appropriate clinic and biochemistry, and imaging.
* Written informed consent
* Speak and understand Danish

Exclusion Criteria (patients and control persons):

* Clinical manifest hepatic encephalopathy
* Consumption of psychoactive substances within 6 days of test
* Organic brain disease (i.e. prior stroke, dementia)
* Hypothyroidism
* Renal failure (creatinine> 150 mg / dL)
* Hyponatremia (Na <125 mmol / L)
* Sepsis or bleeding within one week prior to testing.
* Serious sleep disorders
* Current treatment with lactulose, rifaximin or BCAA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Continuous Reaction Time Method versus Portosystemic Encephalopathy Test | baseline and 3 months
  The investigators are evaluating if the CRT and PSE test are in accordance at inclusion and after 3 months of treatment.

SECONDARY OUTCOMES:
Change in Continuous Reaction Time Method versus Quality of Life (QoL) | baseline and 3 months
  The results from both CRT and PSE test will be compared to the out come of the SF-36 and the SIP (Sickness impact profile) QoL measurements.
Correlation between CRT test and PSE test at inclusion | at baseline
  The investigators wish to evaluate the correlation between the CRT and the PSE test at base line.
Correlation between psychometric test results and quality of life af base line | at base line
  The investigators wish to evaluate the correlation between the psychometric test results (CRT test result and PSE test result) and quality of life. The scientific question is which test correlates best to QoL.

OTHER OUTCOMES:
Danish normal values for the PSE test | at base line
  100 normal Danish persons will be tested using the PSE test to establish the Danish norm.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Schaffalitzky de Muckadell, Professor, Study Director — Odense University Hospital; Jeppe Gram, PhD, MD, Study Chair — Esbjerg Hospital - University Hospital of Southern Denmark; Hendrik Vilstrup, Professor, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Hospital of South West Jutland, Esbjerg
  - Odense University Hospital, Odense